CLINICAL TRIAL: NCT04253223
Title: A Phase I/Ib Pilot Study to Determine the Safety and Efficacy of a Human Anti-glucagon Receptor Antibody (REMD-477) in Controlling Severe Hyperglycemia Due to Copanlisib in Patients With Relapsed or Refractory Lymphoma
Brief Title: A Study to Determine Safety and Efficacy of (REMD-477) in Controlling Hyperglycemia Due to Copanlisib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Herbert Lyerly, Professor, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00102920
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Hyperglycemia Drug Induced
Keywords: hyperglycemia; lymphoma; anti-glucagon receptor antibody; glucagon receptor; Volagidemab
MeSH Terms: conditions — Hyperglycemia; Lymphoma | interventions — volagidemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- REMD-477 (Experimental): REMD-477 (human IgG2 anti-glucagon receptor antibody Volagidemab) will be administered as a subcutaneous injection for three weekly doses
  Interventions: Biological: REMD-477

INTERVENTIONS:
Biological: REMD-477 — REMD-477 will be administered as a subcutaneous injection for three weekly doses
  Other Names: Volagidemab

SUMMARY:
REMD-477 (Volagidemab) is a human anti-glucagon receptor antibody. Its proposed mechanism of action in controlling hyperglycemia is by blocking glucagon receptor (GCGR) signaling. In this way, it increases hepatic glucose uptake, decreases hepatic glycogenolysis and gluconeogenesis, increases glycogen synthesis, and ultimately decreases blood glucose levels. This protocol will test the hypotheses that REMD-477 is safe and tolerable in patients with severe hyperglycemia on copanlisib and that it decreases the risk of severe hyperglycemia in patients receiving copanlisib for relapsed refractory lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Relapsed or refractory lymphoma (Grade 1, 2, 3A)
* Received 2 or more prior lines of systemic therapy for lymphoma
* Experienced glucose >250 mg/dL after copanlisib infusion for treatment of lymphoma

Exclusion Criteria:

* Evidence of histologic transformation
* Follicular Lymphoma Grade 3B
* Active CNS involvement by malignancy
* Elevated AST or ALT > 5x ULN at Screening
* Unmanageable sensitivity to mammalian-derived drug preparations, or to humanized or human antibodies; managed sensitivities to agents such as obinutuzumab or rituximab or similar agents are not exclusionary
* History of drug or alcohol abuse within the last 6 months
* History or family history of pancreatic neuroendocrine tumors or multiple endocrine neoplasia
* History or family history of pheochromocytoma
* Other gastrointestinal, cardiac, renal and CNS (i.e. hypoglycemia unawareness) conditions specific to diabetes that would pose additional risk to subject's safety or interfere with the study evaluation, procedures or completion in the opinion of the treating physician.
* Female subject is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 22 days
  Evaluate the safety of REMD-477 in patients with hyperglycemia due to a PI3 kinase inhibitor
Serious Adverse Events | 22 days
  Evaluate the safety of REMD-477 in patients with hyperglycemia due to a PI3 kinase
Liver Function Tests (LFT) units per liter (u/L) | 22 days
  Evaluate the safety of REMD-477 in patients with hyperglycemia due to a PI3 kinase
Blood Glucose measurements | 22 days
  Evaluate the safety of REMD-477 in patients with hyperglycemia due to a PI3 kinase
Pulse beats per minute | 22 days
  Evaluate the safety of REMD-477 in patients with hyperglycemia due to a PI3 kinase
breathing Rate breaths per minute | 22 days
  Evaluate the safety of REMD-477 in patients with hyperglycemia due to a PI3 kinase

SECONDARY OUTCOMES:
Fasting Glucose levels | 22 days
  Determine efficacy of REMD-477 in preventing copanlisib induced hyperglycemia
Insulin levels | 22 days
  Determine efficacy of REMD-477 in preventing copanlisib induced hyperglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No